CLINICAL TRIAL: NCT00563212
Title: A Pilot Study of Aerosol Interferon-gamma for Treatment of Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Stony Brook University (Other); Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9583; IFB 9583; NCT00212563 (obsolete NCT alias)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Fibrosis
Keywords: Lung Diseases, Interstitial; Fibrosis; Interferons; Pulmonary Fibrosis; Pathologic Processes; Lung Diseases; Fibrosing alveolitis; Interferon-gamma, Recombinant; Aerosols
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Fibrosis; Pathologic Processes; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: aerosol interferon-gamma

INTERVENTIONS:
Drug: aerosol interferon-gamma — aerosol interferon-gamma-1b 100mcg given via nebulizer three times weekly for one year

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a progressive disease for which there is no effective treatment. Interferon-gamma is a medication that has been used for other lung diseases to decrease scarring and fibrosis. Studies of interferon-gamma injected under the skin did not show any improvement in survival in patients with IPF. We hypothesize that giving interferon-gamma as a nebulized mist directly into the lungs can affect the immune system in a way that decreases fibrosis.

DETAILED DESCRIPTION:
Patients with mild-to-moderate idiopathic pulmonary fibrosis (IPF) will be enrolled in a phase I study of aerosol interferon-gamma (IFN-γ). Prior to initiation of treatment, patients will undergo CT of the chest, pulmonary function testing, and bronchoscopy with bronchoalveolar lavage. They will also undergo a lung deposition study to determine the lung dose of IFN-γ that will be delivered with each treatment. Patients will then receive aerosol IFN-γ 100mcg delivered three times weekly via nebulizer for one year. Study patients will be followed monthly to monitor potential side effects, vital signs, and progression of IPF symptoms. Labs will be drawn at regular intervals to monitor for side effects and to measure cytokine levels. Bronchoscopy will be performed at the 6 and/or 12 month visit to compare cytokine levels pre-, during, and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IPF based on accepted criteria (see above) within 12 months prior to screening.
* Age 40-75.
* Absence of significant pulmonary hypertension as measured by right heart catheterization (mPAP ≥ 30 mmHG) or echocardiography (RVSP ≥ 50 mmHg).
* FVC ≥ 55% of predicted baseline value at screening; DLCO ≥ 30% predicted.
* PaO2 ≥ 65 mm Hg at rest on room air
* Patient able to understand and willing to sign a written informed consent and willing to comply with all requirements of the study protocol including lung deposition studies.
* Patient fits criteria for research bronchoscopy and is willing to undergo procedure.

Exclusion Criteria:

* Six minute walk distance of < 200 meters.
* Patient unwilling or unable to undergo research bronchoscopy.
* Patient with known life threatening asthma or severe COPD.
* Patient requiring oxygen therapy for maintenance of adequate arterial oxygenation at rest.
* Patient with hypersensitivity to study medication or other component medication.
* Patient with known severe cardiac disease, severe peripheral vascular disease or seizure disorder which may be exacerbated by study drug administration (contraindications to drug administration as per package insert).
* Pregnant or lactating; Females of child-bearing potential will be required to have negative pregnancy test and be required to use accepted form of birth control (abstinence for study duration is the preferred method).
* Evidence of active infection within one week prior to treatment.
* Any condition, other than IPF, which is likely to result in the death of the patient within one year from study enrollment.
* Abnormal serum laboratory values including:
* Liver function above specified limits: total bilirubin > 1.5 X upper limits of normal, alanine amino transferase > 3X upper limit of normal, alkaline phosphatase > 3X upper limit of normal, albumin < 3.0 at screening.
* CBC outside specified limits: WBC < 2,500/mm3, hematocrit < 30 or > 59, platelets < 100,000/mm3.
* Creatinine > 1.5X upper limits normal at screening.
* Drugs for therapy for pulmonary fibrosis, including corticosteroids, azathioprine and/or cyclophosphamide, or n-acetylcysteine within the previous six weeks.
* Prior therapy with any class of interferon medication.
* Investigational therapy for any indication within the last 28 days.
* In a pulmonary rehabilitation program or planning to attend a pulmonary rehabilitation program.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
safety, tolerability | one year

SECONDARY OUTCOMES:
lung deposition of aerosolized IFN, bronchoalveolar lavage fluid levels of IFN and fibrotic cytokines pre-and post-treatment, pulmonary function testing trends during treatment, descriptive data regarding symptoms and clinical findings | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rany Condos, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- Division of Pulmonary & Critical Care Medicine, NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Goldyn SR, Smaldone GC, Rom WN, Condos R. Safety Profile of Aerosol Interferon-gamma. Abstract submitted to American Thoracic Society for presentation at ATS annual meeting May 2008, Toronto.
- [Derived] Xue Y, Reddy SK, Garza LA. Toward Understanding Wound Immunology for High-Fidelity Skin Regeneration. Cold Spring Harb Perspect Biol. 2022 Jul 1;14(7):a041241. doi: 10.1101/cshperspect.a041241. PMID 35667792